CLINICAL TRIAL: NCT02954913
Title: Simultaneous RESEction of Colorectal Cancer With Synchronous Liver MeTastases (RESECT): A Feasibility Study
Brief Title: Simultaneous Resection of Colorectal Cancer With Synchronous Liver Metastases
Acronym: RESECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Principal Investigator, Pablo Serrano, Hepatobiliary & Pancreatic Surgical Oncologist, Hamilton Health Sciences Corporation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RESECT
Record Dates: First submitted 2016-11-02; First posted 2016-11-04 (Estimated); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: ColoRectal Cancer; Liver Metastases; Liver Metastasis Colon Cancer; Surgery; Complication
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Hepatectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Simultaneous Resection (Experimental): Patients will undergo resection of the colon or rectum and liver in the same anesthetic setting. The type of colorectal and liver resection will be decided by the treating physician. The type of liver resection will be described according to the Couinaud classification and the Brisbane terminology of liver anatomy.
  Interventions: Procedure: Simultaneous Resection

INTERVENTIONS:
Procedure: Simultaneous Resection — Resections of 3 or more segments of the liver will be considered a major liver resection.(Reddy) The anesthetic technique and the order of liver resection or rectal resection will be determined by each surgeon's standards. It is recommended that a low central venous pressure be maintained in order to decrease intraoperative blood loss (Chen; Hughes) and that liver resection be performed prior to colorectal resection in order to keep a low central venous pressure during that part of the case.
  Other Names: Synchronous Colorectal and Liver Resections; Simultaneous Colorectal and Liver Resections; Synchronous Resection

SUMMARY:
Synchronous colorectal cancer with liver metastases, defined as the diagnosis of a primary colorectal tumour and liver metastases within 12 months, is a common problem faced by colorectal and hepatobiliary surgeons.(Adam) The "traditional approach" is to perform staged resections unless the liver resection required is limited (i.e. small wedges of peripheral lesions). The downside of performing staged vs. simultaneous resections is that patients must undergo two major operations instead of one, which limits a patient's ability to return to their pre-surgical state of health in a timely fashion, increasing health care costs (Ejaz) and delaying the start of adjuvant chemotherapy. The disadvantages of a simultaneous approach include longer operating room times potentially increasing the major postoperative complication rate including blood transfusions, surgical site infections, anastomotic leaks and post-hepatectomy liver failure. Recent data from tertiary cancer centres suggest that simultaneous resection of the colon and rectum along with liver resection of any magnitude is feasible and safe.(Silberhumer) Although encouraging, this data comes from specific patients from a highly selected institution, results that are perhaps not generalizable.

This proposal is a feasibility study consisting of a pilot single arm prospective study at two different large-volume Hepatobiliary Centres of patients with synchronous colorectal cancer with liver metastases undergoing simultaneous resection of the colon or rectum and liver to evaluate their complication rates (including the calculation of the comprehensive complication index), quality of life, cost evaluation, and proportion of eligible patients recruited over a 12-month period. The results of this pilot study will provide us with the information necessary to build a large multicentre randomized controlled trial comparing staged vs. simultaneous resection for synchronous colorectal cancer liver metastases.

DETAILED DESCRIPTION:
Approximately 30% of patients with colorectal cancer and liver metastases present with synchronous disease.(Manfredi) Resection of colorectal cancer metastases confined to the liver has been shown to offer long-term survival.(Norlinger; Robertson; Nordlinger) However, the optimal timing of surgical resection of synchronous liver metastases in relation to the primary tumour is not well defined. Prior retrospective cohorts and meta-analyses suggest that the simultaneous approach carries similar postoperative complication and perioperative mortality rates.(Slesser; Yin; Martin; Chua; Feng; Reddy; Jarnagin; Capussotti) Most of these reports however, carry a significant selection bias, as surgeons tend to combine limited liver resections and "straightforward" colorectal resections as opposed to complex resections. Recent studies suggest that the postoperative complication risk is similar even in the case of complex liver resections as well as complex colon resections and rectal cancer resections.(Silberhumer; Vigano) Rectal resections when compared to colon resections are thought to be more complex, due to: a higher risk of anastomotic leakage,(Rullier) the use of specific surgical procedures, such as total mesorectal excision (Heald, MacFarlane) and laparoscopic surgery(Bonjer) and the involvement of a multidisciplinary team to determine the use and timing of neoadjuvant chemoradiotherapy.(Jeong; Kapiteijn) The conclusion of these studies was that further data from prospective randomized studies is needed in order to determine whether simultaneous resection is efficient and safe. Improvements in anesthesia, critical care and surgical resection techniques for both liver and colorectal surgery have enabled innovative surgeons and institutions to perform simultaneous resections in complex liver and colorectal cases in a safe manner, and the simultaneous approach has been adopted by many surgeons despite the lack of studies with rigorous methodology to provide good quality data.

Simultaneous colorectal and liver resection has the potential advantage to decrease the total number of complications following surgery, avoiding a second operation thereby improving patient's quality of life, decreasing overall health care costs and avoiding delays in the administration of postoperative chemotherapy. Although the total number of complications can be reduced by performing a single operation, the operating room time is higher which could lead to a higher proportion of major postoperative complications due to hypothermia, prolonged hypovolemia and higher blood loss.

The decision to perform simultaneous resection varies greatly between surgeons and institutions, with some institutions mostly performing simultaneous resections, to others that only perform staged resection and others that perform a combination of staged and simultaneous resections depending on patients' and tumour characteristics, usually performing larger and more complex resections in a staged approach. There is certainly no standard approach to this problem and it continues to be a topic of debate amongst surgeons, medical oncologists and radiation oncologists.

The investigators propose to undertake a feasibility study, including a prospective single arm trial of patients with synchronous colorectal cancer and liver metastases undergoing simultaneous resection to provide us with important information to prepare a large randomized controlled study of simultaneous vs. staged resection. This feasibility study will provide valuable data on the type and proportion of postoperative complications at 90 days following surgery as measured by the comprehensive complication index(Slankamenac 2013) which will help us better understand the postoperative complication rate of the simultaneous approach and also calculate a sample size for a randomized controlled trial based on this primary outcome. This study will also help define the population that should be included in such a trial (all liver resections vs. only major liver resections, etc.). Set criteria for success of this feasibility study will be clearly stated in this proposal in order to determine if it is possible and ethical to move forward with a larger trial. The results of this study could lead to changes in surgical practice by introducing an innovative approach to treat this disease, in a way that could improve patient's quality of life by decreasing postoperative complications and the number of surgical procedures and at the same time lead to cost savings to the health care system.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who present with resectable synchronous colorectal adenocarcinoma and liver metastases.
2. Patients who have a planned resection of their colorectal adenocarcinoma and liver metastases.
3. Patients who are able to provide informed consent.

Note: The primary tumour or the liver metastases may require neoadjuvant therapy to become resectable. Patients with the following histology are eligible for the study: adenocarcinoma, adenosquamous carcinoma, mixed adenocarcinoma-neuroendocrine tumour (adenocarcinoma with neuroendocrine differentiation). Patients with suspicious colorectal mass with probably liver metastases in which pathology only shows high grade dysplasia are also eligible as long as a liver resection is contemplated as part of the operative plan.

Exclusion Criteria:

1. Extrahepatic disease other than lung.
2. Tumours treated with local transanal excision (patients undergoing transanal total mesorectal excision are eligible).
3. Patients who require a two stage liver resection, prior liver resection.
4. Pregnant or lactating female
5. Absolute contraindications for general anesthesia
6. Patients who require a complex multi-organ pelvic resection, i.e. pelvic exenteration: including bladder, female or male reproductive organs; patients who only require resection of another pelvic organ (including bladder or female reproductive organs or prostate and seminal vesicles) are eligible.
7. Patients undergoing urgent resection of the primary tumour due to bleeding or obstruction in which a simultaneous liver resection is not planned are not eligible for the study, patients who undergo diverting stoma (loop ileostomy or colostomy) prior to resection are eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2017-02-14 (Actual); Primary Completion 2020-03-05 (Actual); Study Completion 2021-02-09 (Actual)

PRIMARY OUTCOMES:
Comprehensive Complication Index | 90 days from the Index Operation
  Postoperative complications used to calculate the Comprehensive Complication Index will be recorded during and following each patient's hospital stay up to 90 days from the index operation and classified according to Clavien-Dindo.(Slankamenac 2013; Dindo; Slankamenac 2014)

SECONDARY OUTCOMES:
Perioperative Mortality | 90 days from the Index Operation
  3.10.2.1. The proportion with its 95% CI of patients who die at 90 days or during the hospital stay for the index operation (perioperative mortality) will be calculated.
Accrual Rate | 12 months from the study's start date
  3.10.2.2. The proportion of eligible patients enrolled in the study over a 12-month period and the proportion of patients who complete the colorectal resection will be assessed.
Global Health-Related Quality of Life | Baseline to 3 months following index surgery
  QoL will be measured using the EORTC-QLQ-C30 (Aaronson; Groenvold) instrument and will be administered at baseline, at 1 and 3 months following surgery.
Cost Analysis | 90 days from the Index Operation
  Health Resource Utilization forms will be used at each patient assessment to determine the number of health related hospital, emergency department or clinic visits, physician appointments and imaging performed. A costing model will be performed by including all factors that drive cost in this patient population.

CONTACTS AND LOCATIONS:
Overall Officials: Pablo E Serrano Aybar, MD, MPH, MSc, FACS, Principal Investigator — Hamilton Health Sciences Corporation
Locations (2):
- Canada (2):
  - Juravinski Hospital and Cancer Centre, Hamilton, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adam R, de Gramont A, Figueras J, Kokudo N, Kunstlinger F, Loyer E, Poston G, Rougier P, Rubbia-Brandt L, Sobrero A, Teh C, Tejpar S, Van Cutsem E, Vauthey JN, Pahlman L; of the EGOSLIM (Expert Group on OncoSurgery management of LIver Metastases) group. Managing synchronous liver metastases from colorectal cancer: a multidisciplinary international consensus. Cancer Treat Rev. 2015 Nov;41(9):729-41. doi: 10.1016/j.ctrv.2015.06.006. Epub 2015 Jun 30. PMID 26417845
- [Background] Ejaz A, Semenov E, Spolverato G, Kim Y, Tanner D, Hundt J, Pawlik TM. Synchronous primary colorectal and liver metastasis: impact of operative approach on clinical outcomes and hospital charges. HPB (Oxford). 2014 Dec;16(12):1117-26. doi: 10.1111/hpb.12302. Epub 2014 Jun 26. PMID 24965845
- [Background] Silberhumer GR, Paty PB, Temple LK, Araujo RL, Denton B, Gonen M, Nash GM, Allen PJ, DeMatteo RP, Guillem J, Weiser MR, D'Angelica MI, Jarnagin WR, Wong DW, Fong Y. Simultaneous resection for rectal cancer with synchronous liver metastasis is a safe procedure. Am J Surg. 2015 Jun;209(6):935-42. doi: 10.1016/j.amjsurg.2014.09.024. Epub 2014 Dec 13. PMID 25601556
- [Background] Manfredi S, Lepage C, Hatem C, Coatmeur O, Faivre J, Bouvier AM. Epidemiology and management of liver metastases from colorectal cancer. Ann Surg. 2006 Aug;244(2):254-9. doi: 10.1097/01.sla.0000217629.94941.cf. PMID 16858188
- [Background] Nordlinger B, Sorbye H, Glimelius B, Poston GJ, Schlag PM, Rougier P, Bechstein WO, Primrose JN, Walpole ET, Finch-Jones M, Jaeck D, Mirza D, Parks RW, Mauer M, Tanis E, Van Cutsem E, Scheithauer W, Gruenberger T; EORTC Gastro-Intestinal Tract Cancer Group; Cancer Research UK; Arbeitsgruppe Lebermetastasen und-tumoren in der Chirurgischen Arbeitsgemeinschaft Onkologie (ALM-CAO); Australasian Gastro-Intestinal Trials Group (AGITG); Federation Francophone de Cancerologie Digestive (FFCD). Perioperative FOLFOX4 chemotherapy and surgery versus surgery alone for resectable liver metastases from colorectal cancer (EORTC 40983): long-term results of a randomised, controlled, phase 3 trial. Lancet Oncol. 2013 Nov;14(12):1208-15. doi: 10.1016/S1470-2045(13)70447-9. Epub 2013 Oct 11. PMID 24120480
- [Background] Robertson DJ, Stukel TA, Gottlieb DJ, Sutherland JM, Fisher ES. Survival after hepatic resection of colorectal cancer metastases: a national experience. Cancer. 2009 Feb 15;115(4):752-9. doi: 10.1002/cncr.24081. PMID 19130462
- [Background] Nordlinger B, Sorbye H, Glimelius B, Poston GJ, Schlag PM, Rougier P, Bechstein WO, Primrose JN, Walpole ET, Finch-Jones M, Jaeck D, Mirza D, Parks RW, Collette L, Praet M, Bethe U, Van Cutsem E, Scheithauer W, Gruenberger T; EORTC Gastro-Intestinal Tract Cancer Group; Cancer Research UK; Arbeitsgruppe Lebermetastasen und-tumoren in der Chirurgischen Arbeitsgemeinschaft Onkologie (ALM-CAO); Australasian Gastro-Intestinal Trials Group (AGITG); Federation Francophone de Cancerologie Digestive (FFCD). Perioperative chemotherapy with FOLFOX4 and surgery versus surgery alone for resectable liver metastases from colorectal cancer (EORTC Intergroup trial 40983): a randomised controlled trial. Lancet. 2008 Mar 22;371(9617):1007-16. doi: 10.1016/S0140-6736(08)60455-9. PMID 18358928
- [Background] Slesser AA, Simillis C, Goldin R, Brown G, Mudan S, Tekkis PP. A meta-analysis comparing simultaneous versus delayed resections in patients with synchronous colorectal liver metastases. Surg Oncol. 2013 Mar;22(1):36-47. doi: 10.1016/j.suronc.2012.11.002. Epub 2012 Dec 14. PMID 23253399
- [Background] Yin Z, Liu C, Chen Y, Bai Y, Shang C, Yin R, Yin D, Wang J. Timing of hepatectomy in resectable synchronous colorectal liver metastases (SCRLM): Simultaneous or delayed? Hepatology. 2013 Jun;57(6):2346-57. doi: 10.1002/hep.26283. PMID 23359206
- [Background] Martin R, Paty P, Fong Y, Grace A, Cohen A, DeMatteo R, Jarnagin W, Blumgart L. Simultaneous liver and colorectal resections are safe for synchronous colorectal liver metastasis. J Am Coll Surg. 2003 Aug;197(2):233-41; discussion 241-2. doi: 10.1016/S1072-7515(03)00390-9. PMID 12892803
- [Background] Chua HK, Sondenaa K, Tsiotos GG, Larson DR, Wolff BG, Nagorney DM. Concurrent vs. staged colectomy and hepatectomy for primary colorectal cancer with synchronous hepatic metastases. Dis Colon Rectum. 2004 Aug;47(8):1310-6. doi: 10.1007/s10350-004-0586-z. PMID 15484344
- [Background] Feng Q, Wei Y, Zhu D, Ye L, Lin Q, Li W, Qin X, Lyu M, Xu J. Timing of hepatectomy for resectable synchronous colorectal liver metastases: for whom simultaneous resection is more suitable--a meta-analysis. PLoS One. 2014 Aug 5;9(8):e104348. doi: 10.1371/journal.pone.0104348. eCollection 2014. PMID 25093337
- [Background] Reddy SK, Pawlik TM, Zorzi D, Gleisner AL, Ribero D, Assumpcao L, Barbas AS, Abdalla EK, Choti MA, Vauthey JN, Ludwig KA, Mantyh CR, Morse MA, Clary BM. Simultaneous resections of colorectal cancer and synchronous liver metastases: a multi-institutional analysis. Ann Surg Oncol. 2007 Dec;14(12):3481-91. doi: 10.1245/s10434-007-9522-5. Epub 2007 Sep 1. PMID 17805933
- [Background] Jarnagin WR, Gonen M, Fong Y, DeMatteo RP, Ben-Porat L, Little S, Corvera C, Weber S, Blumgart LH. Improvement in perioperative outcome after hepatic resection: analysis of 1,803 consecutive cases over the past decade. Ann Surg. 2002 Oct;236(4):397-406; discussion 406-7. doi: 10.1097/01.SLA.0000029003.66466.B3. PMID 12368667
- [Background] Capussotti L, Ferrero A, Vigano L, Ribero D, Lo Tesoriere R, Polastri R. Major liver resections synchronous with colorectal surgery. Ann Surg Oncol. 2007 Jan;14(1):195-201. doi: 10.1245/s10434-006-9055-3. PMID 17080238
- [Background] Rullier E, Laurent C, Garrelon JL, Michel P, Saric J, Parneix M. Risk factors for anastomotic leakage after resection of rectal cancer. Br J Surg. 1998 Mar;85(3):355-8. doi: 10.1046/j.1365-2168.1998.00615.x. PMID 9529492
- [Background] Heald RJ, Ryall RD. Recurrence and survival after total mesorectal excision for rectal cancer. Lancet. 1986 Jun 28;1(8496):1479-82. doi: 10.1016/s0140-6736(86)91510-2. PMID 2425199
- [Background] MacFarlane JK, Ryall RD, Heald RJ. Mesorectal excision for rectal cancer. Lancet. 1993 Feb 20;341(8843):457-60. doi: 10.1016/0140-6736(93)90207-w. PMID 8094488
- [Background] Bonjer HJ, Deijen CL, Abis GA, Cuesta MA, van der Pas MH, de Lange-de Klerk ES, Lacy AM, Bemelman WA, Andersson J, Angenete E, Rosenberg J, Fuerst A, Haglind E; COLOR II Study Group. A randomized trial of laparoscopic versus open surgery for rectal cancer. N Engl J Med. 2015 Apr 2;372(14):1324-32. doi: 10.1056/NEJMoa1414882. PMID 25830422
- [Background] Jeong SY, Park JW, Nam BH, Kim S, Kang SB, Lim SB, Choi HS, Kim DW, Chang HJ, Kim DY, Jung KH, Kim TY, Kang GH, Chie EK, Kim SY, Sohn DK, Kim DH, Kim JS, Lee HS, Kim JH, Oh JH. Open versus laparoscopic surgery for mid-rectal or low-rectal cancer after neoadjuvant chemoradiotherapy (COREAN trial): survival outcomes of an open-label, non-inferiority, randomised controlled trial. Lancet Oncol. 2014 Jun;15(7):767-74. doi: 10.1016/S1470-2045(14)70205-0. Epub 2014 May 15. PMID 24837215
- [Background] Kapiteijn E, Marijnen CA, Nagtegaal ID, Putter H, Steup WH, Wiggers T, Rutten HJ, Pahlman L, Glimelius B, van Krieken JH, Leer JW, van de Velde CJ; Dutch Colorectal Cancer Group. Preoperative radiotherapy combined with total mesorectal excision for resectable rectal cancer. N Engl J Med. 2001 Aug 30;345(9):638-46. doi: 10.1056/NEJMoa010580. PMID 11547717
- [Background] Slankamenac K, Graf R, Barkun J, Puhan MA, Clavien PA. The comprehensive complication index: a novel continuous scale to measure surgical morbidity. Ann Surg. 2013 Jul;258(1):1-7. doi: 10.1097/SLA.0b013e318296c732. PMID 23728278
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Background] Fong Y, Fortner J, Sun RL, Brennan MF, Blumgart LH. Clinical score for predicting recurrence after hepatic resection for metastatic colorectal cancer: analysis of 1001 consecutive cases. Ann Surg. 1999 Sep;230(3):309-18; discussion 318-21. doi: 10.1097/00000658-199909000-00004. PMID 10493478
- [Background] Bismuth H. Revisiting liver anatomy and terminology of hepatectomies. Ann Surg. 2013 Mar;257(3):383-6. doi: 10.1097/SLA.0b013e31827f171f. PMID 23386236
- [Background] Strasberg SM. Nomenclature of hepatic anatomy and resections: a review of the Brisbane 2000 system. J Hepatobiliary Pancreat Surg. 2005;12(5):351-5. doi: 10.1007/s00534-005-0999-7. PMID 16258801
- [Background] Chen H, Merchant NB, Didolkar MS. Hepatic resection using intermittent vascular inflow occlusion and low central venous pressure anesthesia improves morbidity and mortality. J Gastrointest Surg. 2000 Mar-Apr;4(2):162-7. doi: 10.1016/s1091-255x(00)80052-9. PMID 10675239
- [Background] Hughes MJ, Ventham NT, Harrison EM, Wigmore SJ. Central venous pressure and liver resection: a systematic review and meta-analysis. HPB (Oxford). 2015 Oct;17(10):863-71. doi: 10.1111/hpb.12462. Epub 2015 Aug 20. PMID 26292655
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Slankamenac K, Nederlof N, Pessaux P, de Jonge J, Wijnhoven BP, Breitenstein S, Oberkofler CE, Graf R, Puhan MA, Clavien PA. The comprehensive complication index: a novel and more sensitive endpoint for assessing outcome and reducing sample size in randomized controlled trials. Ann Surg. 2014 Nov;260(5):757-62; discussion 762-3. doi: 10.1097/SLA.0000000000000948. PMID 25379846
- [Background] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Background] Groenvold M, Klee MC, Sprangers MA, Aaronson NK. Validation of the EORTC QLQ-C30 quality of life questionnaire through combined qualitative and quantitative assessment of patient-observer agreement. J Clin Epidemiol. 1997 Apr;50(4):441-50. doi: 10.1016/s0895-4356(96)00428-3. PMID 9179103
- [Derived] Serrano PE, Gafni A, Parpia S, Ruo L, Simunovic M, Meyers BM, Reiter H, Wei A, Gallinger S, Karanicolas P, Hallet J, Devaud N, Levine M. Simultaneous resection of colorectal cancer with synchronous liver metastases (RESECT), a pilot study. Int J Surg Protoc. 2018 Feb 1;8:1-6. doi: 10.1016/j.isjp.2018.01.001. eCollection 2018. PMID 31851740